CLINICAL TRIAL: NCT06491550
Title: A Phase I Randomized, Single-blind, Placebo-controlled, and Sequential Group Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD4144 Following Single and Multiple Ascending Doses Via Intravenous Administration, and an Open-label, 2-Period, 2-Sequence, Cross-over Study to Assess the Effects of Intravenous AZD4144 on Rosuvastatin and Furosemide Pharmacokinetics in Healthy Participants
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD4144 as Well as the Impact of AZD4144 on the Pharmacokinetics of Rosuvastatin and Furosemide in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: D9440C00002
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Healthy Participants
Keywords: Pharmacokinetic (PK); Pharmacodynamic (PD); Drug-drug interaction (DDI); Single ascending dose (SAD); Multiple ascending dose (MAD)
MeSH Terms: interventions — Rosuvastatin Calcium; Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (17):
- Part A1-Cohort 1 (Experimental): Participants will receive one single ascending dose of AZD4144.
  Interventions: Drug: AZD4144- Part A
- Part A1- Cohort 2 (Experimental): Participants will receive one single ascending dose of AZD4144.
  Interventions: Drug: AZD4144- Part A
- Part A1-Cohort 3 (Experimental): Participants will receive one single ascending dose of AZD4144.
  Interventions: Drug: AZD4144- Part A
- Part A2-Japanese cohort 1 (Experimental): Participants will receive one single ascending dose of AZD4144.
  Interventions: Drug: AZD4144- Part A
- Part A2: Japanese Cohort 2 (Experimental): Participants will receive one single ascending dose of AZD4144.
  Interventions: Drug: AZD4144- Part A
- Part A3-Chinese Cohort (Experimental): Participants will receive one single ascending dose of AZD4144.
  Interventions: Drug: AZD4144- Part A
- Part B1- Cohort 1 (Experimental): Participants will receive multiple ascending doses of AZD4144.
  Interventions: Drug: AZD4144- Part B
- Part B1- Cohort 2 (Experimental): Participants will receive multiple ascending doses of AZD4144.
  Interventions: Drug: AZD4144- Part B
- Part B1- Cohort 3 (Experimental): Participants will receive multiple ascending doses of AZD4144.
  Interventions: Drug: AZD4144- Part B
- Part B2- Japanese Cohort (Experimental): Participants will receive multiple ascending doses of AZD4144.
  Interventions: Drug: AZD4144- Part B
- Part C Cohort- Treatment C1 (Experimental): Participants will receive rosuvastatin and furosemide.
  Interventions: Drug: Rosuvastatin and Furosemide- Part C
- Part C cohort- Treatment C2 (Experimental): Participants will receive rosuvastatin, furosemide, and AZD4144.
  Interventions: Drug: Rosuvastatin, Furosemide, and AZD4144 Part C
- Part A1- Placebo (Placebo Comparator): Participants will receive matching placebo.
  Interventions: Drug: Placebo- Part A
- Part A2- Placebo (Placebo Comparator): Participants will receive matching placebo.
  Interventions: Drug: Placebo- Part A
- Part A3- Placebo (Placebo Comparator): Participants will receive matching Placebo.
  Interventions: Drug: Placebo- Part A
- Part B1- Placebo (Placebo Comparator): Participants will receive matching Placebo.
  Interventions: Drug: Placebo- Part B
- Part B2- Placebo (Placebo Comparator): Participants will receive matching Placebo.
  Interventions: Drug: Placebo- Part B

INTERVENTIONS:
Drug: AZD4144- Part A — Part A: Participants will be administered a single dose of AZD4144 on Day 1 via Intravenous (IV) infusion.
  Arms: Part A1- Cohort 2; Part A1-Cohort 1; Part A1-Cohort 3; Part A2-Japanese cohort 1; Part A2: Japanese Cohort 2; Part A3-Chinese Cohort
Drug: Placebo- Part A — Part A: Participants will be administered a single dose of placebo on Day 1 via IV infusion.
  Arms: Part A1- Placebo; Part A2- Placebo; Part A3- Placebo
Drug: AZD4144- Part B — Part B: Participants will be administered a single dose of AZD4144 on Day 1 and Day 12 via IV infusion.
  Participants will be administered multiple doses of AZD4144 from Day 4 to Day 11 via IV infusion.
  Arms: Part B1- Cohort 1; Part B1- Cohort 2; Part B1- Cohort 3; Part B2- Japanese Cohort
Drug: Placebo- Part B — Part B: Participants will be administered a single dose of placebo on Day 1 and Day 12via IV infusion. Participants will be administered multiple doses of placebo from Day 4 to Day 11 via IV infusion.
  Arms: Part B1- Placebo; Part B2- Placebo
Drug: Rosuvastatin and Furosemide- Part C — Participants will be administered a single oral dose of 10 mg Rosuvastatin and 1 mg Furosemide.
  Arms: Part C Cohort- Treatment C1
Drug: Rosuvastatin, Furosemide, and AZD4144 Part C — Participants will be administered a single oral dose of 10 mg Rosuvastatin, 1 mg Furosemide and a single dose of AZD4144 via IV infusion.
  Arms: Part C cohort- Treatment C2

SUMMARY:
This study consists of 3 parts: Part A, Part B and Part C. This study will compare the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of AZD4144 with placebo in healthy participants, in Part A and Part B. Part C of this study will investigate the possibility of drug-drug interaction (DDI) between IV AZD4144 and oral rosuvastatin and furosemide by evaluating the PK of rosuvastatin and furosemide when administered alone and in combination with single IV dose of AZD4144

DETAILED DESCRIPTION:
This is a Phase I, randomized study in healthy participants and consists of 3 parts; Part A, Part B and Part C. Part A and B are single-blind, placebo-controlled with single ascending dose (SAD) and multiple ascending dose (MAD) sequential group design, respectively. Part C is an open-label, 2-period, 2-sequence, cross-over design study. Part A and B of the study will assess the safety, tolerability, PK, and PD of AZD4144 solution for infusion compared with placebo while Part C will investigate the possibility of DDI between IV AZD4144 and oral rosuvastatin and furosemide by evaluating the PK of rosuvastatin and furosemide when administered alone and in combination with single IV dose of AZD4144

The study will comprise of:

* A screening period of maximum 28 days.
* A residential period which lasts from,

  * Day -1 to Day 4 (single dose on Day 1) for Part A
  * Day -1 to Day 15 (dosed on days 1, 4-12) for Part B
  * Day -1 to Day 3 (dose on Day 1) and Day 9 to Day 12 (dose on Day 10) for Part C
* A final follow-up visit,

  * On Day 10+3 for Part A
  * On Day 20+3 for Part B and C

ELIGIBILITY:
Inclusion Criteria:

* All females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit.
* Females of childbearing potential must not be lactating and if heterosexually active must agree to use an approved method of highly effective contraception.
* Females of non-childbearing potential must be confirmed at the Screening Visit.
* Sexually active fertile male participants with partners of childbearing potential must adhere to the contraception methods.
* Have a BMI between 18 and 32 kg/m2 inclusive at both Screening and Admission and weigh at least 45 kg at Screening.
* For healthy Japanese cohorts (Part A2 and Part B2): healthy male and female participants are to be Japanese, defined as having both parents and 4 grandparents who are Japanese. This includes second and third generation participants of Japanese descent whose parents or grandparents are living in a country other than Japan.
* For healthy Chinese cohort (Part A3): healthy male and female Chinese participants for whom both parents and all grandparents are Chinese and not lived outside of China for more than 10 years.

Exclusion Criteria:

* History of any clinically important disease or disorder or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure, or trauma.
* Clinically significant serious active and chronic infections.
* Any history or evidence of TB (active or latent).
* Known history of primary immunodeficiency (congenital or acquired) or an underlying condition that predisposes to infection.
* Bacillus Calmette Guérin vaccine within one year prior to signing the ICF.
* Any abnormal laboratory values at the Screening Visit or on Admission to the Clinical Unit.
* Any positive result on Screening for serum Hepatitis B surface antigen (HBsAg), anti-Hepatitis B core (HBc), hepatitis C antibody, or Human immunodeficiency virus (HIV).
* Any clinically important abnormalities in ECG.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity.
* Known hypersensitivity to furosemide and rosuvastatin (for Part C only)
* History of alcohol abuse or excessive intake of alcohol or current smokers or those who have smoked or used nicotine products.
* Use of drugs with enzyme inducing properties or of any prescribed or nonprescribed medication or of systemic hormonal contraceptives.
* Clinical signs and symptoms consistent with COVID-19.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) (Part A and Part B) | Part A: Day 1 to Day 10+3; Part B: Day 1 to Day 20+3.
  To assess the safety and tolerability of AZD4144 following IV administration of single (Part A) and multiple (Part B) ascending doses in healthy participants.
Area under plasma concentration-time curve from time 0 to infinity (AUCinf) (Part C) | Treatment period 1: Day 1 to 3; Treatment period 2: Day 10 to 12.
  To evaluate the effect of AZD4144 on the PK of rosuvastatin and furosemide in healthy participants.
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) (Part C) | Treatment period 1: Day 1 to 3; Treatment period 2: Day 10 to 12.
  To evaluate the effect of AZD4144 on the PK of rosuvastatin and furosemide in healthy participants.
Maximum observed drug concentration (Cmax) (Part C) | Treatment period 1: Day 1 to 3; Treatment period 2: Day 10 to 12.
  To evaluate the effect of AZD4144 on the PK of rosuvastatin and furosemide in healthy participants.

SECONDARY OUTCOMES:
Cmax (Part A and Part B) | Part A: Day 1 to Day 10+3; Part B: Day 1 to Day 20+3
  To characterize the PK of AZD4144 following IV administration of single (Part A) and multiple (Part B) ascending doses.
AUClast (Part A and Part B) | Part A: Day 1 to Day 10+3; Part B: Day 1 to Day 20+3
  To characterize the PK of AZD4144 following IV administration of single (Part A) and multiple (Part B) ascending doses
AUCinf (Part A) | Part A: Day 1 to Day 10+3
  To characterize the PK of AZD4144 following IV administration of single (Part A) ascending doses.
Area under concentration-time curve in the dosing interval (AUCτ) (Part B only) | Part B: Day 1 to Day 20+3
  To characterize the PK of AZD4144 following IV administration of multiple (Part B) ascending doses
Renal clearance of drug from plasma (CLR) (Part A and Part B) | Part A: Day 1 to 3; Part B: Day 1, 12 and 20+3
  To characterize the PK of AZD4144 following IV administration of single (Part A) and multiple (Part B) ascending doses.
PD analysis: Levels of disease-specific biomarkers (Part A and Part B) | Part A: Day -1 to 4; Part B: Day -1 to Day 1, Day 12 to Day 15
  To assess the effect of AZD4144 on levels of disease-specific biomarkers. (Part A and Part B)
Number of participants with adverse events (AEs) (Part C) | Part C: Day 1 to Day 20+3
  To assess the safety and tolerability of AZD4144 in combination with rosuvastatin and furosemide in healthy participants.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Glendale, California
  - Research Site, Brooklyn, Maryland

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/